CLINICAL TRIAL: NCT02908997
Title: MindMate: A Single Case Experimental Design Study of a Reminder System for People With Mild Dementia
Brief Title: MindMate: A Study of a Reminder System for People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GN16NE538
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 week baseline (Experimental): 5 week baseline data collection followed by 6 week MindMate intervention
  Interventions: Other: MindMate
- 6 week baseline (Experimental): 6 week baseline data collection followed by 6 week MindMate intervention
  Interventions: Other: MindMate
- 7 week baseline (Experimental): 7 week baseline data collection followed by 6 week MindMate intervention
  Interventions: Other: MindMate

INTERVENTIONS:
Other: MindMate — A dementia-specific mobile reminding application

SUMMARY:
A study to investigate the effectiveness of a reminder tool application at increasing performance on memory tasks in people with mild dementia

DETAILED DESCRIPTION:
Background

Memory difficulties are a core feature of dementia. These include difficulties remembering to do something at a specific time and place in the future (Prospective Memory). Although a range of electronic prospective memory aids currently exist (e.g. "Neuropage"), the evidence supporting their use among the dementia population remains limited. "Mindmate" is a recently developed mobile application that aims to support individuals with a diagnosis of dementia, improving self-management skills and quality of life.

Aims

This study will explore the effectiveness of "MindMate" reminder alerts delivered to a smart phone or tablet computer as a memory aid for people with a diagnosis of Mild Dementia.

Method

Three participants with a diagnosis of dementia, who are considered to be in the early stages and who report everyday prospective memory difficulties, will be recruited from Older People Community Mental Health teams within Greater Glasgow and Clyde. The participants will own a smart phone or tablet and will be living with a partner or family member who will also participate in the study. During the initial baseline phase, the partner or family member will monitor the number of pre defined tasks the participant remembered and forgot. The partner or family member will record this information on a weekly monitoring form and this phase will last between five to seven weeks. This will be followed by a five-week intervention phase where "MindMate" reminder alerts will be sent to the participant's phone or tablet. Again, tasks that require remembering will be identified prior to the intervention phase, and family members or carers will monitor their success on a form. Results will be analysed using visual inspection and Tau-U analysis.

Applications

This study will provide information on the effectiveness of a form of assistive technology at supporting people with a dementia, which could improve quality of life of those with a diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* has a diagnosis of Mild Dementia, according to International Classification of Diseases (ICD) 10 Criteria
* has received the diagnosis from a psychiatrist
* owns a smart phone or tablet
* has a family member/partner/carer who is willing to monitor memory aid use
* has capacity to consent to being involved in the research
* is reporting memory difficulties that are affecting them in daily life

Exclusion Criteria:

* visual or auditory difficulties which cannot be corrected through the use of appropriate aids
* has a pre-existing neurological or severe psychiatric problem (e.g. bipolar disorder, psychosis)
* has a diagnosis of dementia that is considered to be in the moderate to severe stages
* those whose first language is not English
* those with a diagnosed or suspected developmental learning disability
* those who are currently using online or electronic memory aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Memory | 6 weeks
  Number of target events the participant remembered to complete

SECONDARY OUTCOMES:
Acceptability | Change from baseline to 6 week post-intervention
  Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, BSc DClinPsy PhD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No